CLINICAL TRIAL: NCT06161376
Title: Prospective Study Evaluating the Role of Urinary Sphingosine 1-Phosphate as a Biomarker for Detrusor Hyperactivity in Multiple Sclerosis
Brief Title: Role of Urinary Sphingosine 1-Phosphate as a Biomarker for Detrusor Hyperactivity in Multiple Sclerosis
Acronym: SEP-1
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/23/0346
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urinary test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- multiple sclerosis: Patients diagnosed with MS requiring urodynamic assessment will be recruited during outpatient visits at Toulouse University Hospital. Initial consultations will involve questionnaire completion, 72-hour voiding diaries, and urine sample collection just before urodynamic assessments.
  Interventions: Other: S1P level

INTERVENTIONS:
Other: S1P level — Patients will undergo urinary S1P level assessments before treatment, 6 weeks post-injection, and following any symptomatic changes that may lead to another urodynamic assessments.

SUMMARY:
This study aims to establish a link between urinary Sphingosine 1-Phosphate (S1P) levels and detrusor activity in multiple sclerosis (MS) patients. MS often involves urological symptoms, primarily overactive bladder. The gold standard for evaluation and treatment monitoring is invasive urodynamic testing. Preliminary research at Toulouse University Hospital suggests urinary S1P levels may be a potential biomarker for detrusor activity in MS. This study aims to confirm this potential biomarker's utility.

ELIGIBILITY:
Inclusion Criteria:

* French residents enrolled in the social security system
* Patients diagnosed with multiple sclerosis (according to McDonald 2017 criteria), whether receiving treatment or not
* Patients scheduled for urodynamic assessment as part of their management

Exclusion criteria:

* Pregnant or lactating females
* Patients under legal guardianship
* Untreated urinary tract infection at the time of inclusion
* Known anatomical subvesical obstruction Known pelvic floor disorder Urothelial carcinoma Interstitial cystitis Augmentation cystoplasty

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with multiple sclerosis
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
S1P concentration | Day 0, after 6 months
  To compare of the urinary concentration of S1P related to creatinine in urine sample, as a function of the detrusor activity determined at BUD, before and after a first intra-detrusor injection of botulinum toxin.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Game, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Toulouse Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No